CLINICAL TRIAL: NCT02982473
Title: Registry of Malignant Arrhythmias and Sudden Cardiac Death - Influence of Diagnostics and Interventions
Acronym: RACE-IT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Michael Behnes, Sub-PI, Universitätsmedizin Mannheim
Other Study IDs: 2016-612N-MA
Record Dates: First submitted 2016-11-29; First posted 2016-12-05 (Estimated); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Ventricular Tachycardia; Ventricular Fibrillation; Sudden Cardiac Death; Coronary Angiography; Electrophysiologic Testing (EP); Catheter Ablation; Percutaneous Coronary Intervention (PCI); Internal Cardioverter Defibrillator (ICD)
MeSH Terms: conditions — Tachycardia, Ventricular; Ventricular Fibrillation; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The "Registry of Malignant Arrhythmias and Sudden Cardiac Death - Influence of Diagnostics and Interventions (RACE-IT)" represents a mono-centric registry of patients being hospitalized suffering from malignant arrythmias (ventricular tachycardia or fibrillation) and sudden cardiac death (SCD).

Detailed findings of patients' clinical outcome regarding mortality and co-morbidities related to the presence of invasive diagnostics or therapies including coronary angiography, percutaneous coronary intervention (PCI), electrophysiological testing (EP), catheter ablation and implanted cardiac devices (e.g. implantable cardioverter-defibrillators) will be documented. Patients will be included when being hospitalized from the year 2004 until today.

ELIGIBILITY:
Inclusion Criteria:

Hospitalization due to:

* ventricular tachycardia
* ventricular fibrillation
* sudden cardiac death

Exclusion Criteria:

* not diagnosed with one or more of the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being hospitalized with diagnoses of ventricular tachycardia, ventricular fibrillation and/or sudden cardiac death at the First Department of Medicine, University Medical Centre Mannheim, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of ventricular arrythmias (i.e. ventricular fibrillation, ventricular tachykardia, asystole, SCD) | Through study completion, potentially up to 12 years, depending on patient inclusion/first event and patients lifetime

SECONDARY OUTCOMES:
Incidence of coronary artery disease (CAD) and PCI in patients with VF/VT/SCD | Through study completion, potentially up to 12 years, depending on patient inclusion/first event and patients lifetime
Incidence of invasive electrophysiologic testing (EP) and catheter ablation | Through study completion, potentially up to 12 years, depending on patient inclusion/first event and patients lifetime
Incidence of treatment with cardiac devices (i.e. ICD, CCM, CRT-D) | Through study completion, potentially up to 12 years, depending on patient inclusion/first event and patients lifetime
Incidences of recurrent malignant tachycardias, all-cause mortality, arrhythmia-related death, re-PCI/ACVB, re-ablation, further therapy with cardiac devices | Through study completion, potentially up to 12 years, depending on patient inclusion/first event and patients lifetime

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Akin, Prof. Dr., Principal Investigator — First Deparment of Medicine, University Medical Centre Mannheim (UMM), Germany; Theodor-Kutzer-Ufer 1-3; 61867 Mannheim, Germany
Locations (1):
- First Department of Medicine, University Medical Centre Mannheim, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Weidner K, Behnes M, Schupp T, Hoppner J, El-Battrawy I, Ansari U, Saleh A, Taton G, Reiser L, Bollow A, Reichelt T, Ellguth D, Engelke N, Bertsch T, Grosse Meininghaus D, Hoffmann U, Akin I. Cardiac disease and prognosis associated with ventricular tachyarrhythmias in young adults and adults. BMC Cardiovasc Disord. 2022 Mar 31;22(1):136. doi: 10.1186/s12872-022-02552-6. PMID 35361107
- [Derived] Rusnak J, Behnes M, Schupp T, Lang S, Reiser L, Taton G, Bollow A, Reichelt T, Ellguth D, Engelke N, Ansari U, El-Battrawy I, Bertsch T, Nienaber CA, Akin M, Mashayekhi K, Weiss C, Borggrefe M, Akin I. Statin therapy is associated with improved survival in patients with ventricular tachyarrhythmias. Lipids Health Dis. 2019 May 24;18(1):119. doi: 10.1186/s12944-019-1011-x. PMID 31122256
- [Derived] Schupp T, Behnes M, Weiss C, Nienaber C, Lang S, Reiser L, Bollow A, Taton G, Reichelt T, Ellguth D, Engelke N, Ansari U, El-Battrawy I, Bertsch T, Akin M, Mashayekhi K, Borggrefe M, Akin I. Beta-Blockers and ACE Inhibitors Are Associated with Improved Survival Secondary to Ventricular Tachyarrhythmia. Cardiovasc Drugs Ther. 2018 Aug;32(4):353-363. doi: 10.1007/s10557-018-6812-z. PMID 30074111